CLINICAL TRIAL: NCT04451161
Title: A Hybrid Type 2 Trial of Trauma-Focused Cognitive Behavioral Therapy and a Pragmatic Individual-Level Implementation Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Minnesota (Other)
Responsible Party: Principal Investigator, Aaron Lyon, Associate Professor, School of Medicine: Psychiatry: Childrens Division, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00008401; 1R01MH119148-01A1 (NIH)
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Evidence-Based Practices; CBT; School Health Services; Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma | interventions — Schools; Therapeutics

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The care provider is not masked to the intervention condition they are in (ie, TF-CBT vs TAU), but will be masked to the implementation strategy (ie, Attention Control vs. BASIS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BASIS with TF-CBT (Other): Implementation intervention: experimental arm (Beliefs and Attitudes for Successful Implementation in Schools)
  Clinical Intervention: experimental arm (Trauma-Focused CBT)
  Interventions: Behavioral: Beliefs and Attitudes for Successful Implementation in Schools (BASIS); Behavioral: Trauma-Focused Cognitive-Behavioral Therapy
- Attention Control (AC) with TF-CBT (Other): Implementation intervention: control arm
  Clinical Intervention: experimental arm (Trauma-Focused CBT)
  Interventions: Behavioral: Trauma-Focused Cognitive-Behavioral Therapy; Behavioral: Attention Control
- Enhanced Treatment as Usual (Other): Implementation intervention: non-applicable
  Clinical Intervention: control arm (Enhanced TAU)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Beliefs and Attitudes for Successful Implementation in Schools (BASIS) — BASIS blended (i.e., multifaceted and protocolized) implementation strategy, which occurs at the beginning of active implementation. BASIS is designed to facilitate observable implementation outcomes, including EBP adoption and intervention fidelity, via strategic education, motivational Interviewing, and social influence strategies.
  Arms: BASIS with TF-CBT
Behavioral: Trauma-Focused Cognitive-Behavioral Therapy — TF-CBT is an evidence-based treatment that helps children from elementary to high school to address the negative effects of trauma and promote greater emotion and behavior regulation, including processing their traumatic memories, overcoming problematic thoughts and behaviors, and developing effective coping and interpersonal skills. It also includes a treatment component for parents or other caregivers. Parents can learn skills related to stress management, positive parenting, behavior management, and effective communication.
  Arms: Attention Control (AC) with TF-CBT; BASIS with TF-CBT
Behavioral: Treatment as Usual — Scaffolded intervention as usual. Includes: initial assessment of trauma symptoms, psychoeducation, follow-up planning and support.
  Arms: Enhanced Treatment as Usual
Behavioral: Attention Control — Didactic presentation of implementation-related content (e.g., information about the importance of implementing, definitions of key terms, etc.) to control for facilitator, dose, information provided, and delivery platform
  Arms: Attention Control (AC) with TF-CBT

SUMMARY:
This research project is a hybrid type 2 effectiveness-implementation trial that simultaneously examines (1) the effectiveness of a trauma-focused intervention for youth in the education sector and (2) the impact of a theory-driven pragmatic implementation strategy designed to increase the adoption, fidelity, and sustainment of evidence-based treatments (EBTs). This trial will include 120 clinicians and 480 students, and it is designed to test the cost effectiveness and impact of Trauma-Focused Cognitive Behavioral Therapy (TF-CBT) in a new setting that increases access to mental health care - schools (Aim 1); test the cost effectiveness, immediate impact, and sustained impact of the Beliefs and Attitudes for Successful Implementation in Schools (BASIS) implementation strategy on proximal mechanisms and implementation outcomes (Aims 2a, 2b, 2d); and conduct sequential mixed-methods data collection to explain residuals (i.e., clinicians whose implementation behavior is unaccounted for by the mediation model) (Aim 2c).

ELIGIBILITY:
Clinicians will be included if they (a) provide school-based services in a participating district; (b) have not previously received formal training in TF-CBT; and (c) are not actively receiving support to implement another trauma-focused intervention.

Students subjects will meet TF-CBT eligibility criteria, including (a) be within the TF-CBT developmental range (ages 8 to 19), (b) have traumatic event exposure (e.g., exposure to violence), and (c) significant post-traumatic stress symptoms.

Ages: 7 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Lyon, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Lyon AR, Pullmann MD, Dorsey S, Levin C, Gaias LM, Brewer SK, Larson M, Corbin CM, Davis C, Muse I, Joshi M, Reyes R, Jungbluth NJ, Barrett R, Hong D, Gomez MD, Cook CR. Protocol for a hybrid type 2 cluster randomized trial of trauma-focused cognitive behavioral therapy and a pragmatic individual-level implementation strategy. Implement Sci. 2021 Jan 7;16(1):3. doi: 10.1186/s13012-020-01064-1. PMID 33413511

RESULTS

PARTICIPANT FLOW:
Recruitment Details: School districts across the United States were recruited to participate in the study, where the district leaders provided a list of potential eligible clinicians currently employed in schools in the district. The eligibility criteria for clinicians were a) provided school-based services for the participating school district; b) did not receive formal training in TF-CBT or CBT+; c) did not receive support to implement another trauma-focused intervention.
Groups:
- BASIS With TF-CBT (Provider): Participants who received training for the implementation intervention BASIS and the clinical intervention, trauma-focused CBT.
- AC (Attention Control) With TF-CBT (Provider): Participants who received control for the implementation intervention and training for trauma-focused CBT for clinical intervention.
- Enhanced Treatment as Usual (Provider): Participants who received control for both implementation and clinical intervention.
- BASIS With TF-CBT (Students): Students recruited by providers who received training for the interventions: implementation (BASIS) and clinical (TF-CBT).
- AC (Attention Control) With TF-CBT (Student): Students recruited by providers who received control for the implementation intervention and training for TF-CBT for clinical intervention.
- Enhanced Treatment as Usual (Student): Students recruited by providers who received control for both implementation and clinical intervention.
Period: Overall Study
Arm/Group | BASIS With TF-CBT (Provider) | AC (Attention Control) With TF-CBT (Provider) | Enhanced Treatment as Usual (Provider) | BASIS With TF-CBT (Students) | AC (Attention Control) With TF-CBT (Student) | Enhanced Treatment as Usual (Student)
Started | 62 | 65 | 64 | 34 | 32 | 35
End of Training Period (Provider) | 47 | 45 | 54 | 0 | 0 | 0
End of Active Phase of the Study (Provider) | 37 | 30 | 48 | 0 | 0 | 0
3-month Follow up (Student) | 0 | 0 | 0 | 26 | 24 | 21
Completed | 31 | 28 | 42 | 21 | 19 | 17
Not Completed | 31 | 37 | 22 | 13 | 13 | 18
Not completed — Lost to Follow-up | 28 | 37 | 22 | 13 | 11 | 14
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The eligibility criteria for clinicians: a) provided school-based services for the participating school district; b) did not receive formal training in TF-CBT or CBT+; c) did not receive support to implement another trauma-focused intervention.
  Eligible students recruited by participating providers: a) within the TF-CBT development age ( 8-19); b) experienced a traumatic event exposure (e.g., exposure to violence); and c) significant post-traumatic stress symptoms.
Groups:
- Total: Total of all reporting groups
Arm/Group | BASIS With TF-CBT (Provider) | AC (Attention Control) With TF-CBT (Provider) | Enhanced Treatment as Usual (Provider) | BASIS With TF-CBT (Students) | AC (Attention Control) With TF-CBT (Student) | Enhanced Treatment as Usual (Student) | Total
Number analyzed (Participants) | 62 | 65 | 64 | 34 | 32 | 35 | 292
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 34 | 32 | 35 | 101
  Between 18 and 65 years | 62 | 64 | 63 | 0 | 0 | 0 | 189
  >=65 years | 0 | 1 | 1 | 0 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Students were recruited by providers who participated in the study. The students needed to be a) within the TF-CBT development range (age 8-19), b) experienced a traumatic event (e.g., exposure to violence), and c) have significant post-traumatic stress symptoms. Only categorical age was collected for provider participants; therefore, the mean and standard deviation cannot be calculated.
  Years
    number analyzed (Participants) | 0 | 0 | 0 | 34 | 32 | 35 | 101
    (all) |  |  |  | 11 (2.7) | 12 (3.2) | 11.2 (2.5) | 11.4 (2.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 58 | 58 | 60 | 16 | 14 | 17 | 223
  Male | 2 | 6 | 4 | 18 | 12 | 16 | 58
  Transgender | 0 | 0 | 0 | 0 | 2 | 1 | 3
  Non-binary | 2 | 0 | 0 | 0 | 2 | 1 | 5
  Unknown or not reported | 0 | 1 | 0 | 0 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 10 | 3 | 1 | 20
  Not Hispanic or Latino | 59 | 63 | 63 | 24 | 28 | 34 | 271
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 1 | 1 | 4 | 1 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 2 | 0 | 1 | 4
  Black or African American | 2 | 2 | 3 | 0 | 2 | 2 | 11
  White | 55 | 55 | 55 | 14 | 17 | 23 | 219
  More than one race | 2 | 2 | 1 | 13 | 8 | 5 | 31
  Unknown or Not Reported | 2 | 4 | 1 | 3 | 5 | 3 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62 | 65 | 64 | 34 | 32 | 35 | 292

OUTCOME MEASURES:

1. Primary Outcome: TF-CBT Adoption and Penetration
Description: Participants provided data every 2-3 months for up to two years, reporting:
  How many students received CPSS-V (PTSD screener)? With how many students was TF-CBT initiated? With how many students was it completed? This allowed for monitoring of both reach (screening) and implementation (initiation/completion) of TF-CBT.
Time Frame: 18 Months- Active phase (timepoint 6 to 9); Sustainment phase (timepoint 10 to 12)
Population: Of the randomized participants, the overall number of participants analyzed was still active after the training period. The measure breaks down the number of providers who administered the screener with at least one student, and then adopted (started or completed) the trauma-informed intervention with at least one student.
Measure: Count of Participants; unit: Participants
Arm/Group | BASIS With TF-CBT (Provider) | AC (Attention Control) With TF-CBT (Provider) | Enhanced Treatment as Usual (Provider)
Number analyzed (Participants) | 47 | 45 | 54
Participants
  Administered CPSS-V with at least one student. | 33 | 26 | 33
  Started TF-CBT with at least one student. | 31 | 26 | 21
  Completed TF-CBT with at least one student. | 11 | 12 | 19
Statistical Analysis 1: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as administered CPSS-V) was binary: either the participant adopted at least one of these components with a student, or they did not at the beginning of the active phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.591, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants administered the CPSS-V to at least one student beginning of the active phase
Statistical Analysis 2: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as administered CPSS-V) was binary: either the participant adopted at least one of these components with a student, or they did not by the end of the active phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.032, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants administered the CPSS-V to at least one student by the end of the active phase
Statistical Analysis 3: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); One of the primary TF-CBT adoption outcomes (defined as administered CPSS-V) was binary: either the participant adopted at least one of these components with a student at the end of the sustainment phase, or they did not. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.054, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants administered the CPSS-V to at least one student by the end of the sustainment phase
Statistical Analysis 4: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as started TF-CBT) was binary: either the participant adopted at least one of these components with a student, or they did not at the beginning of the active phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.98, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants started TF-CBT with at least one student at the beginning of the active phase
Statistical Analysis 5: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as started TF-CBT) was binary: either the participant adopted at least one of these components with a student, or they did not by the end of the active phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.068, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants started TF-CBT with at least one student by the end of the active phase
Statistical Analysis 6: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as started TF-CBT) was binary: either the participant adopted at least one of these components with a student, or they did not by the end of the sustainment phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.165, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants started TF-CBT with at least one student by the end of the sustainment phase
Statistical Analysis 7: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as completed TF-CBT) was binary: either the participant adopted at least one of these components with a student, or they did not by the end of the active phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.191, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants completed TF-CBT with at least one student by the end of the active phase
Statistical Analysis 8: Comparison: BASIS With TF-CBT (Provider) vs AC (Attention Control) With TF-CBT (Provider); The primary TF-CBT adoption outcome (defined as completed TF-CBT) was binary: either the participant adopted at least one of these components with a student, or they did not by the end of the sustainment phase. A chi-squared test was used as a superiority test to determine whether participants in the BASIS group had higher TF-CBT adoption rates compared to the Attention Control group; Test type: Superiority; p = 0.86, Chi-squared — We performed a chi-squared analysis comparing the study groups (BASIS vs. Attention Control) on whether participants completed TF-CBT with at least one student at the end of the sustainment phase

2. Primary Outcome: Child PTSD Symptom Scale for DSM-V
Description: The Child PTSD Symptom Scale Self-Report for DSM-5 (CPSS-V) is a modified version of the original CPSS-SR adapted for DSM-5 criteria. The scale includes 20 PTSD symptom items scored on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("6 or more times a week / severe"), where higher scores indicate greater symptom severity. The scale includes 7 functioning items rated as "yes" or "no." The total score ranges from 0 to 80, with higher scores reflecting worse PTSD symptom severity.
Time Frame: 6 Months - Baseline (T1); 3-month follow up (T2); 6-month follow up (T3)
Population: All the participants (students) who received trauma-informed intervention- TF-CBT or Enhanced treatment as usual.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- BASIS With TF-CBT (Student): Students recruited by providers who received training for the interventions: implementation (BASIS) and clinical (TF-CBT).
- Attention Control With TF-CBT (Student): Students recruited by providers who received control for the implementation intervention and training for TF-CBT for clinical intervention.
Arm/Group | BASIS With TF-CBT (Student) | Attention Control With TF-CBT (Student) | Enhanced Treatment as Usual (Student)
Number analyzed (Participants) | 34 | 32 | 35
Score on a scale
  Baseline (T1) | 34.7 (15.9) | 39.3 (18.7) | 37.1 (16.1)
  3-month follow up (T2): number analyzed (Participants) | 26 | 24 | 21
  3-month follow up (T2) | 28.3 (16.2) | 34.4 (16.2) | 28.1 (17.4)
  6-month follow up (T3): number analyzed (Participants) | 21 | 19 | 17
  6-month follow up (T3) | 26.1 (17.7) | 32.2 (18.8) | 19.4 (16.3)
Statistical Analysis 1: Comparison: BASIS With TF-CBT (Student) vs Enhanced Treatment as Usual (Student); We compared the BASIS group (receiving TF-CBT) against Enhanced Treatment as Usual to evaluate whether TF-CBT reduced trauma-related PTSD symptoms over time, as measured by CPSS-V scores (higher scores indicate greater symptom severity); Test type: Superiority; p = 0.22, Mixed Models Analysis — Mixed model analysis was used (students were clustered under the providers who recruited them) to understand if BASIS+TF-CBT has a greater effect on decreasing trauma PTSD symptoms (measured using CPSS-V) over time; Slope = 3.425, 95% CI 2-sided [-2.064 to 8.915], Standard Error of Mean 2.783
Statistical Analysis 2: Comparison: Attention Control With TF-CBT (Student) vs Enhanced Treatment as Usual (Student); We compared the AC group (receiving TF-CBT) against Enhanced Treatment as Usual to evaluate whether TF-CBT reduced trauma-related PTSD symptoms over time, as measured by CPSS-V scores (higher scores indicate greater symptom severity); Test type: Superiority; p = 0.075, Mixed Models Analysis — Mixed model analysis was used (the students were clustered under the providers who recruited them) to understand if AC+TF-CBT has a greater effect on decreasing trauma PTSD symptoms (measured using CPSS-V) over time; Slope = 4.97, 95% CI 2-sided [-.502 to 10.443], Standard Error of Mean 2.774

3. Primary Outcome: Mood and Feelings Questionnaire - Short
Description: The Short Mood and Feelings Questionnaire (SMFQ) is a 13-item self-report measure assessing recent emotional and behavioral states. It consists of descriptive phrases rated based on how often they applied to the subject over the past two weeks: 0 ("not at all"), 1 ("sometimes"), or 2 ("most of the time"). The total score ranges from 0 to 26, with higher scores indicating greater severity of depressive symptoms (worse outcome).
Time Frame: 6 Months - Baseline (T1); 3-month follow up (T2); 6-month follow up (T3)
Population: All the participants (students) who received trauma-informed intervention- TF-CBT or Enhanced Treatment as Usual.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BASIS With TF-CBT (Student) | Attention Control With TF-CBT (Student) | Enhanced Treatment as Usual (Student)
Number analyzed (Participants) | 34 | 32 | 35
score on a scale
  Baseline (T1) | 10.3 (7.7) | 11.7 (7.1) | 10.7 (5.9)
  3-month follow up (T2): number analyzed (Participants) | 26 | 24 | 21
  3-month follow up (T2) | 7.7 (4.8) | 12.1 (6.3) | 7.2 (4.4)
  6-month follow-up (T3): number analyzed (Participants) | 21 | 19 | 17
  6-month follow-up (T3) | 6.8 (6.3) | 10 (7.3) | 4.9 (4.3)
Statistical Analysis 1: Comparison: BASIS With TF-CBT (Student) vs Enhanced Treatment as Usual (Student); We compared the BASIS group (receiving TF-CBT) against Enhanced Treatment as Usual to evaluate whether TF-CBT decreased children's negative moods and feelings due to their trauma (higher score indicates more negative mood and feelings); Test type: Superiority; p = 0.284, Mixed Models Analysis — Mixed model analysis was used (students were clustered under the providers who recruited them) to understand if BASIS+TF-CBT has a greater effect on decreasing negative mood and feelings symptoms (measured using SMFQ) over time; Slope = 1.024, 95% CI 2-sided [-.855 to 2.904], Standard Error of Mean .952
Statistical Analysis 2: Comparison: Attention Control With TF-CBT (Student) vs Enhanced Treatment as Usual (Student); We compared the AC group (receiving TF-CBT) against Enhanced Treatment as Usual to evaluate whether TF-CBT decreased children's negative moods and feelings due to their trauma (higher score indicates more negative mood and feelings); Test type: Superiority; p = .046, Mixed Models Analysis — Mixed model analysis was used (students were clustered under the providers who recruited them) to understand if AC+TF-CBT has a greater effect on decreasing negative mood and feelings symptoms (measured using SMFQ) over time; Slope = 1.908, 95% CI 2-sided [.03 to 3.786], Standard Error of Mean .951

ADVERSE EVENTS:
Time Frame: 6 months- Baseline (T1), 3-month follow up (T2), 6-month follow up (T3)
Description: Any adverse events (including serious ones) were only collected for students (none collected for providers). Identified through a CPSS-V item assessing self-harm (other adverse event). If a student scored >0 ('not at all') on this item, the protocol followed:
  Notifying the school mental health provider (provider participant) and the parent (with the student's consent). Based on the severity, escalating to the on-call study clinician to develop a safety plan.
Arm/Group | BASIS With TF-CBT (Student) | Attention Control With TF-CBT (Student) | Enhanced Treatment as Usual (Student) | BASIS With TF-CBT (Provider) | AC (Attention Control) With TF-CBT (Provider) | Enhanced Treatment as Usual (Provider)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 0/35 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/32 | 0/35 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 3/34 | 4/32 | 2/35 | 0/0 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BASIS With TF-CBT (Student) (N=34) | Attention Control With TF-CBT (Student) (N=32) | Enhanced Treatment as Usual (Student) (N=35) | BASIS With TF-CBT (Provider) (N=0) | AC (Attention Control) With TF-CBT (Provider) (N=0) | Enhanced Treatment as Usual (Provider) (N=0)
Suicidal Ideation/ Self-harm (Social circumstances) | 3 (3) | 4 (4) | 2 (2) | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT04451161/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT04451161/ICF_001.pdf